CLINICAL TRIAL: NCT01109368
Title: The Rogosin Institute Homozygous Familial Hypercholesterolemia Repository
Status: Recruiting | Type: Observational
Sponsor: The Rogosin Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 0912010770
Record Dates: First submitted 2010-04-21; First posted 2010-04-23 (Estimated); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Homozygous Familial Hypercholesterolemia
Keywords: Autosomal Dominant Familial Hypercholesterolemia
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, monocytes
Oversight: Data Monitoring Committee: No

SUMMARY:
This repository will establish for the first time a system to carefully assess and monitor over time the general health and the amount of cholesterol in the arteries of U.S. children and adults with homozygous familial hypercholesterolemia (hoFH). Patients with this very rare disorder have very high blood levels of cholesterol from birth due to the inheritance of an abnormal gene from each parent. As a result, if untreated, heart attacks and sudden death occur in childhood. Treatments such as LDL-apheresis and liver transplant will lower the cholesterol level, but the best treatment and the best way to monitor the effect of the treatment on the arteries are unknown. The collection of clinical data and blood for analysis of known and yet-to-be discovered markers and predictors of arterial disease will yield new information about the natural history of the disorder and response to treatment. The repository will greatly aid the development of specific protocols that seek to learn more about this disease and new therapies.

DETAILED DESCRIPTION:
Detailed information of "standard of care" procedures will be compiled in a database. These include medical history and physical exam, lipid profiles and other standard blood tests, dietary evaluation and counseling, cardiology evaluation including EKG and echocardiogram,ultrasound of carotids and femoral arteries, CT angiogram and, if indicated, intracoronary angiography (ICA) with intravascular ultrasound (IVUS) and stress echo or nuclear stress testing.

The recommendation for treatment will be individualized. Current options are a) FDA approved cholesterol-lowering medications: statins, ezetimibe b) LDL-apheresis c) liver transplant d) portacaval shunt e) investigational drugs. Treatment of vascular and/or valvular disease may include aspirin, beta blockers, clopidogrel, angioplasty with metal stent, coronary artery bypass surgery, aortic valve repair/replacement.

Research procedures will include medical photos of skin xanthomas, blood assays (apolipoproteins A and B, LDL particle size, homocysteine, TNF, IL-6, insulin, glucose, ICAM, VCAM, P and E selectin, and endothelial progenitor cells), and DNA analysis of the genes for the LDL receptor and other lipid-related genes.

ELIGIBILITY:
Inclusion criteria:

1. Patients of any age and sex who meet clinical or genetic criteria for hoFH as follows:

* Documented, untreated fasting LDL cholesterol level of > 500 mg/dL and triglycerides < 200 mg/dL on a cholesterol-lowering diet for at least 8 weeks with secondary causes excluded, AND:

  * DNA confirmation of a double mutation of the LDL receptor or apoB gene OR
  * LDL > 160 mg/dL in both biological parents not associated with a disorder know to elevate LDL OR
  * Coronary artery disease in one or both parents or grandparents < 55 years for males, < 65 for females OR
  * Tendinous/cutaneous xanthomas < age 10 or coronary artery disease < age 20

Exclusion criteria:

1. Inability of patient, or, if less than 18, a parent, to sign informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Males and females of any age with severely elevated LDL cholesterol levels without secondary causes and a family history consistent with an autosomal dominant disorder.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2010-06 (Actual); Primary Completion 2030-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Change in disease progression | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Lisa C. Hudgins, M.D., Principal Investigator — The Rogosin Institute
Locations (1):
- The Rogosin Institute, Weill Cornell Medical College, New York, New York, United States